CLINICAL TRIAL: NCT03338166
Title: Role of LDH as a Predictor of Treatment Outcomes in Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nourhan Yousef, Principal Investigator, Assiut University
Other Study IDs: URL
Record Dates: First submitted 2017-06-17; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: Patients with Hepatocellular carcinoma who treated with sorafenib and measure LDH serum level one month pre and post treatment
  Interventions: Other: LDH serum level
- Group B: Patients with Hepatocellular carcinoma who treated with trans catheter arterial chemo embolization (TACE) and measure LDH serum level one month pre and post treatment
  Interventions: Other: LDH serum level
- Group C: Patients with Hepatocellular carcinoma who treated surgically and measure LDH serum level one month pre and post treatment
  Interventions: Other: LDH serum level
- Group D: Patients with Hepatocellular carcinoma who don't receive treatment and asses LDH serum level for 3months
  Interventions: Other: LDH serum level

INTERVENTIONS:
Other: LDH serum level — Blood sample to measure LDH as a predictor of Hepatocellular carcinoma treatment outcome

SUMMARY:
Hepatocellular carcinoma represents the commonest primary cancer of the liver.serum lactate dehydrogenase is an indirect marker of tumor hypoxia,angioneogenesis and worse prognosis.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) represents the commonest primary cancer of the liver. Incidence is increasing and HCC has risen to become the 5th commonest malignancy worldwide and the third leading cause of cancer related death, exceeded only by cancers of the lung and stomach. HCC prevalence is higher in sub-Saharan Africa, central and Southeast Asia.Serum lactate dehydrogenase (LDH) levels is an indirect marker of tumor hypoxia, angioneogenesis and worse prognosis. Lactic dehydrogenase (LDH), which is a glycolytic enzyme, composed of four polypeptide chains, each one encoded by separate gene (M and H), exists in various types of human tissue and neoplasms. LDH is a key enzyme in the conversion pyruvate to lactate under anaerobic conditions .Five isoforms of LDH have been identified as a result of the five different combinations of polypeptide subunits.

Hypoxia represents a clinical biological mechanism for treatment resistance in cancer cells via the formation of new blood vessels. Furthermore, a growing body of evidence indicates that hypoxia might actually promote cancer development.

ELIGIBILITY:
Inclusion Criteria:

* patients with Hepatocellular carcinoma diagnosed by biopsy or imaging criteria and alpha feto protein.
* signed informed consent before registration in study
* Eastern Cooperative oncology Groups Performance status between 0 and 2.

Exclusion Criteria:

* Cachexia or poor condition
* pregnant or human chorionic gonadotropin positive
* patient with another liver tumor
* Any previous treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients resident at oncology department at luxor international hospital who diagnosed as apatient with Hepatocellular carcinoma
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-02 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
serum LDH level as a predictor of response in hepatocellular carcinoma | 2 months
  To evaluate if serum LDH level can be used as a predictor of response in patients receiving different lines of treatment for hepatocellular carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Aml R Ibrahim, Lecturer, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided